CLINICAL TRIAL: NCT04643327
Title: Double-blind Randomised-controlled Within-subject Crossover Trial to Determine Levetiracetam Efficacy for Memory Impairment in Parkinson's Disease: A Proof-of-concept Study
Brief Title: Uncovering a Novel Therapeutic Target to Reduce Dementia Risk in Parkinson's Disease
Acronym: TRIP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Queensland University of Technology (Other); Johns Hopkins University (Other); Cleveland Clinic Lou Ruvo Center for Brain Health (Unknown); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Principal Investigator, Nadeeka Dissanyaka, NHMRC Boosting Dementia Research Leadership Fellow, The University of Queensland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC/2020/QRBW/69379
Record Dates: First submitted 2020-11-18; First posted 2020-11-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Mild Cognitive Impairment; Memory Impairment
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction; Memory Disorders | interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: Double-blind randomised-controlled within-subject crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): 125mg Levetiracetam capsules taken twice daily (morning and evening) for 14 days
  Interventions: Drug: Levetiracetam
- Placebo arm (Placebo Comparator): 125mg maize starch-based placebo capsules taken twice daily (morning and evening) for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam — Levetiracetam is currently approved in Australia and the U.S.A. for epilepsy. We will be providing levetiracetam in capsule form, 125mg levetiracetam in each capsule.
  Arms: Active arm
Drug: Placebo — Placebo intervention will be maize-starch filled capsules with identical physical features to the active capsules.
  Arms: Placebo arm

SUMMARY:
The present study is a proof-of-concept clinical trial to test the efficacy of low doses of a repurposed anti-epileptic drug (levetiracetam) in treating memory problems in Parkinson's disease (PD). Neuroimaging techniques will be used to determine the effect of the drug on specific brain regions (hippocampal subfields). Finally, baseline brain activity of PD patients with memory problems will be compared to PD patients without memory problems and healthy older adults to determine if activity in specific brain regions (hippocampal subfields) can be used to predict memory problems in PD. This information will be useful for future clinical trials to target drugs to these brain regions.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease patients with amnestic Mild Cognitive Impairment
* Parkinson's Disease patients with no memory impairment
* Healthy volunteers
* All participants must be eligible to take MRI scans

Exclusion Criteria:

* Dementia
* Contraindication to having MRI
* Bipolar disorder, Schizophrenia, Alcohol or substance abuse
* Major depression
* Suicidal Ideation
* Difficulty complying with protocol requirements
* Significant non-PD neurological disease
* Vascular dementia
* Sensitivity to levetiracetam
* Use of anticonvulsant medications
* Use of other excluded medications
* Severe renal impairment
* Clinically significant abnormalities in B12 or thyroid function test (below normative range for elderly)
* Females of childbearing potential

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pattern separation performance (behavioural outcome) | Immediately after 2 weeks of treatment
  Participants' behavioural performance on the pattern separation fMRI paradigm, as measured by their proportionate accuracy of identifying the critical "lure" trials.
Hippocampal DG/CA3 subfield activity | Immediately after 2 weeks of treatment
  Participants' brain activation during the pattern separation fMRI paradigm, as measured by their activation in the critical dentate gyrus (DG)/CA3 subfield of the hippocampus during the critical "lure" trials of the pattern separation task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Queensland Centre for Clinical Research, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] Dissanayaka N, Pourzinal D, Byrne GJ, Yang J, McMahon KL, Pontone GM, O'Sullivan JD, Adam R, Littleford R, Chatfield M, Lehn A, Mari Z, Bakker A. Levetiracetam for the treatment of mild cognitive impairment in Parkinson's disease: a double-blind controlled proof-of-concept trial protocol. Pilot Feasibility Stud. 2023 Nov 22;9(1):189. doi: 10.1186/s40814-023-01406-y. PMID 37993889